CLINICAL TRIAL: NCT03997253
Title: Optimizing Long-term Survival in Organ Transplantation: From Physiopathology to Optimized Patient Management
Acronym: BIOSUPORT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Collaborators: University Hospital Federation FHU SUPORT (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 87RI18-0027
Record Dates: First submitted 2019-06-24; First posted 2019-06-25 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Organ Transplantation
Keywords: organ transplantation, graft, biological collection.
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: various blood and urine samples will be collected from the recipient at D0, D1, D3, D7, D14, M1, M3, M6 and M12 and intraoperative bile collection ancillary studies : stools at D0 D7 M1 and M3 will be collected for liver transplant patient
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- blood, bile and urine samples (Experimental): blood and urine samples at D0,D1, D3 D7, D14, M1, M3, M6 and M12
  Interventions: Other: blood and urine samples

INTERVENTIONS:
Other: blood and urine samples — various blood and urine samples will be collected from the recipient at D0, D7, D14, M1, M3, M6 and M12 and intraoperative bile collection

SUMMARY:
Increased indications for transplantation continue to worsen the shortage of organs and need the extension of graft sampling criteria and the search for new potential sources of organs. Despite undeniable success in the short term, due to major advances in surgery, medicine and research, transplant recipients continue to face the risk of chronic rejection and long-term complications.

The University Hospital Federation "FHU SUPORT" was created to optimize the chances of success of the organ transplant and improve the quality of life of the transplanted patient. FHU SUPORT 's ambition is based on a translational strategy that presents two priority areas:

Axis 1: Optimization, evaluation, conditioning of the donor, graft, recipient Axis 2: Personalized follow-up of the transplanted patient in the short and long term Identifying factors for long-term graft and patient survival through translational research from a common cohort and biological collection will predict transplant rejection, prolong graft function, or improve the patient's care.

ELIGIBILITY:
Inclusion Criteria:

* Male or female over 18 (no age limit)
* affiliated to a social security organization
* Recipient (s) of a kidney, liver or heart transplant
* followed by at least one of the FHU SUPORT centers (Tours, Poitiers, Limoges, Rennes)
* having given informed consent to participate in the cohort.

Exclusion Criteria:

* Patient unable to understand the information given by the investigator
* People under the protection of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Estimated)
Dates: Start 2020-12-21 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Survival of the graft | 12 months

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Limoges hospital, Limoges
  - Poitiers Hospital, Poitiers
  - Rennes Hospital, Rennes
  - Tours hospital, Tours

IPD SHARING:
Plan to Share IPD: No